CLINICAL TRIAL: NCT04339504
Title: Long-term Follow-up Study of Safety and Explore Efficacy in Subjects Who Completed SMUP-IA-01 Phase Ⅰ Clinical Trial
Brief Title: Follow-up Safety and Efficacy Evaluation on Subjects Who Completed Phase I Clinical Trial
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medipost Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-SMUP-IA-P01-F/U
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Knee Osteoarthritis
Keywords: human umbilical cord blood derived mesenchymal stem cells; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SMUP-IA-01(low-dose) (Experimental): A single knee administration of SMUP-IA-01 (low-dose, 4.0 x 10^6 cells/2mL) (2 ml of 1% sodium hyaluronate injection is administered before administration of SMUP-IA-01)
  Interventions: Biological: SMUP-IA-01(low-dose)
- SMUP-IA-01(mid-dose) (Experimental): A single knee administration of SMUP-IA-01 (mid-dose, 1.0 x 10^7 cells/2mL) (2 ml of 1% sodium hyaluronate injection is administered before administration of SMUP-IA-01)
  Interventions: Biological: SMUP-IA-01(mid-dose)
- SMUP-IA-01(high-dose) (Experimental): A single knee administration of SMUP-IA-01 (high-dose, 2.0 x 10^7 cells/2mL) (2 ml of 1% sodium hyaluronate injection is administered before administration of SMUP-IA-01)
  Interventions: Biological: SMUP-IA-01(high-dose)

INTERVENTIONS:
Biological: SMUP-IA-01(low-dose) — A single knee administration of SMUP-IA-01(low-dose, 4.0 x 10^6 cells/2mL)
  Other Names: Human umbilical cord blood-derived mesenchymal stem cells
  Arms: SMUP-IA-01(low-dose)
Biological: SMUP-IA-01(mid-dose) — A single knee administration of SMUP-IA-01(mid-dose, 1.0 x 10^7 cells/2mL)
  Other Names: Human umbilical cord blood-derived mesenchymal stem cells
  Arms: SMUP-IA-01(mid-dose)
Biological: SMUP-IA-01(high-dose) — A single knee administration of SMUP-IA-01(high-dose, 2.0 x 10^7 cells/2mL)
  Arms: SMUP-IA-01(high-dose)

SUMMARY:
This is a follow-up study to investigate the long-term safety and explore efficacy of SMUP-IA-01, for the treatment of Knee Osteoarthritis. Subjects who participated in and completed the initial stage of the Phase I trial (NCT04037345 ) will be followed-up until 60 months.

DETAILED DESCRIPTION:
The subjects will be followed up at 6-month, 12-month, 24-month, 36-month, 48-month and 60-month after the initial administration of SMUP-IA-01.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who completed the safety and explore efficacy evaluations in SMUP-IA-01 Phase I clinical trial.
2. Subjects who have been treated with either SMUP-IA-01 at least 6 months ago.
3. Subjects who voluntarily decided to participate and signed the consent form after receiving explanations on the clinical trial.

Exclusion Criteria:

1. Subjects who were not enrolled in phase 1 clinical trial of SMUP-IA-01 for assessing safety and explore efficacy.
2. Other subjects, excluding those listed above, who were deemed unsuitable by the PI

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-04-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change of total score in WOMAC (Western Ontario and McMaster University) | Month 12, 24, 36, 48 and 60 after treatment
  Comparing WOMAC total score changes with baseline scores of SMUP-IA-01 phase I trial and scores of f/u study at 12 months, 24 months, 36 months, 48 months and 60months after treatment (score range 0-96, higher score represent worse symptoms).

SECONDARY OUTCOMES:
Change of score in WOMAC three subscales (Pain, stiffness, physical function) | Month 12, 24, 36, 48 and 60 after treatment
  The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68).
Change of score in 100 mm VAS (Visual Analogue Scale) | Month 12, 24, 36, 48 and 60 after treatment
  The score ranges from "0" or no pain to "100" very severe pain
Change of score in IKDC(International Knee Documentation Committee) | Month 12, 24, 36, 48 and 60 after treatment
  The scores for each category are summed up and divided into 87, which is the maximum score possible, and then is evaluated by converting it into a scale of 100 points. Higher score indicates better function and less symptoms for the knee.
Change of score in WORMS(Whole-Organ Magnetic Resonance iMaging Score) | Month 12 and 24 after treatment
  For structural and tissue evaluation of knee, MRI image of detailed knee parts are graded from min. 0 to max. 6. Lower number indicate normal status
Change in K&L(Kellgren-Lawrence) grade | Month 12 and 24 after treatment
  The K & L grade is 0 to 4 Grade, which means that the higher the grade, the greater the joint damage and the stenosis of the joint
Change in joint space width | Month 12 and 24 after treatment
  Evaluation of disease progression in target knee as ascertained by change from baseline in joint space width (JSW) determined using radiography
Change in mechanical axis, anatomical axis | Month 12 and 24 after treatment
  The degree of deformation of the lower half of the body is measured by measuring the angles of the mechanical axis and the anatomical axis with respect to the vertical axis. Mechanical axis: A line connecting the femoral head center point and the ankle joint center point. Anatomical axis: The middiaphyseal line of the femur and tibia
Rate of surgery to treat application site after treatment of SMUP-IA-01 | Month 6, 12, 24, 36, 48 and 60 after treatment
  Rate of surgery to treat application site after treatment of SMUP-IA-01
Changes in biomarker | Month 12 after treatment
  Comparing biomarker changes with baseline of SMUP-IA-01 phase I trial and scores of f/u study at 12 months after treatment. urine C-terminal cross-linking telopeptides of collagen type II (CTX II), serum cartilage oligomeric matrix protein (COMP), serum matrix metalloproteinase-3 (MMP-3)

CONTACTS AND LOCATIONS:
Overall Officials: Myungchul LEE, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul national University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No